CLINICAL TRIAL: NCT05200078
Title: Deep Inspiration Breath-hold Radiotherapy for Left-sided Breast Cancer in Reducing Early Cardiac Injury: a Phase II Prospective Study
Brief Title: Deep Inspiration Breath-hold Radiotherapy for Left-sided Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shu lian Wang (Unknown)
Responsible Party: Sponsor-Investigator, Shu lian Wang, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: 2020-2-4023
Record Dates: First submitted 2021-12-13; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer; Cardiac Event
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radiotherapy at free-breathing: breast/chest wall+-RNI 43.5Gy/15f/3w（tumor bed 49.5Gy/15f/3w) delivered at free-breathing
- Radiotherapy at deep inspiration breath-hold: breast/chest wall+-RNI 43.5Gy/15f/3w（tumor bed 49.5Gy/15f/3w) delivered at deep inspiration breath-hold
  Interventions: Device: Deep inspiration breath-hold technique

INTERVENTIONS:
Device: Deep inspiration breath-hold technique — Selective application of deep inspiration breath-hold technique
  Groups: Radiotherapy at deep inspiration breath-hold

SUMMARY:
Postoperative breast radiotherapy (RT) has been associated with increased risk of heart toxicity. However, there is a lack of knowledge for radiation-induced early cardiovascular injury, especially for hypofractionated RT. This study aims to prospectively detect and predict early clinical or subclinical cardiac events in women undergoing adjuvant RT for breast cancer.

DETAILED DESCRIPTION:
Women with left-sided breast cancer undergo hypofractionated RT at either free-breathing or deep inspiration breath-hold. The incidence and potential clinical, dosimetric and biological indicators of early clinical or subclinical cardiac injury are investigate at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Primary left-sided breast cancer post surgery
* Planning for adjuvant breast/chest wall +-RNI

Exclusion Criteria:

* History of cardiovascular disease
* Previous chest radiation
* Bilateral breast cancers

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: women with left-sided breast cancer planning for adjuvant radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinical or subclinical cardiac injury | two years
  predefined cardiac events

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China